CLINICAL TRIAL: NCT03679390
Title: The Effect of Ketamine Between Generations in Operation Theater- Focus on Electroencephalogram Changes
Brief Title: The Electroencephalogram and Clinical Effect of Ketamine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201605031RINC
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2020-06

CONDITIONS: Electroencephalogram; Consciousness, Loss of
MeSH Terms: conditions — Unconsciousness | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Use same medication for different generations, focus on the reactions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10-20 y/o (Experimental): We will include the teenagers who need intravenous general anesthesia(IVGA), and inject propofol with/without ketamine 0.5mg/kg with full monitor. We will record the EEG during the who operation.
  Interventions: Drug: Ketamine
- 20-40y/o group (Experimental): We will include patients who need IVGA, and inject propofol with/without ketamine 0.5mg/kg with full monitor. We will record the EEG during the who operation.
  Interventions: Drug: Ketamine
- >70 y/o (Experimental): We will include patients who need IVGA, and inject propofol with/without ketamine 0.5mg/kg with full monitor. We will record the EEG during the who operation.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — With the Ketamine group, we add ketamine 0.5mg/kg for anesthesia.
  Other Names: control

SUMMARY:
The electroencephalography (EEG) is a noninvasive medical technique for monitoring and recording the electrical activity of brain. The Hilbert-Huang Transformation (HHT) was proposed to decompose EEG signal into intrinsic mode functions (IMF). HHT can obtain instantaneous frequency data and work well for nonstationary and nonlinear data. We applied this method in perioperative EEG signal analysis in order to find the energy shift and quantify the energy change during general anesthesia. Ketamine was a depolarized sedative which was wildly used in anesthesia. We are trying to find the energy change after ketamine injection, and the interaction between different oscillations in EEG. The whole brain mapping for ketamine and other sedatives interaction is the next step.

DETAILED DESCRIPTION:
Method: In the first year, we will record 60 patients who received general anesthesia, their EEG data recorded from bi-spectral index (BIS) monitor. Under the same anesthesia depth, the experimental group use ketamine 0.5mg/kg; while the control group using alfentanil 0.01mg/kg injection. Both perioperative data were recorded included heart rate, blood pressure and surgical time. We decompose the raw EEG data from BIS monitor with EMD, and we observe difference between IMFs, and quantifying energy change. Second year: We will extend the EEG monitor to temporal lobe, parietal lobe and occipital lobe. Besides the whole brain mapping method for detecting energy change after ketamine injection; we also tried to find the interactions between oscillations. Finally, we want to apply the analysis method to pediatric patients, try to find the difference of ketamine reaction between generations. Anticipated Results: We anticipate that we can quantify the energy of EEG by Emperical mode decomposition(EMD), and ketamine injection can cause different energy change with other sedatives. We will find the energy traveling in EEG with EMD decomposition. We will find that HHT is more suitable for EEG analysis in clinical practicing. With the whole brain mapping method, we can understand the electrical activity during general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiology I-II Not allergic to BIS probe Do not have wound or scar over forehead area

Exclusion Criteria:

patient refuse not suitable for propofol or ketamine injection

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Ketamine increase the dissociation energy in EEG | one year
  ANOVA measurement

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided